CLINICAL TRIAL: NCT04797520
Title: Assessing Diagnostic Accuracy of Core Stethoscope Auscultation vs. Point of Care Ultrasound in Localizing Correct Placement of Endotracheal Tube
Brief Title: Diagnostic Accuracy of Core Stethoscope Auscultation vs. Point of Care Ultrasound in Placement of Endotracheal Tube
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 60429
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Intubation Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Other): All participants will have placement of ETT confirmed using both Core stethoscope and point-of-care ultrasound
  Interventions: Device: Eko CORE Stethoscope; Device: Point of care ultrasound

INTERVENTIONS:
Device: Eko CORE Stethoscope — Eko CORE stethoscope will be used as a visual and auditory means of confirming placement of ETT
Device: Point of care ultrasound — Point of care ultrasound will be used as a means of confirming placement of ETT. This is the "gold standard" used in standard of care

SUMMARY:
Misplacement of endotracheal tube (ETT) can have devastating complications for patients, some of which include respiratory failure, atelectasis, and pneumothorax.

There are a number of ways to verify the correct placement of ETT, with the stethoscope auscultation being commonly used despite its low accuracy (60-65%) in distinguishing tracheal from bronchial intubation (4-6). The gold standard techniques include Chest X Ray or fiberoptic bronchoscope (7-8), with a recent study showing point-of-care ultrasound. However, these techniques are expensive, time-consuming, often not readily available and require substantial training before users can reliably utilize them. Given intubation is often performed in urgent clinical settings, a technique that can reliably yet efficiently localize ETT would be beneficial.

Tele-auscultation system via Core stethoscope (Eko, Berkeley, CA) has been shown to be effective in identifying pathologic heart murmur (10) yet its potential use in guiding the correct placement of ETT has not been explored. We set out to study the suitability of Core stethoscope in detecting the correct placement of ETT.

ELIGIBILITY:
Inclusion Criteria:

* Any patients under the age of 18
* Surgery requiring an ETT
* Consent/parental consent to

Exclusion Criteria:

* Possible difficult airway
* Significant lung pathology
* with any major cardiac anomaly

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Localization of endotracheal tube placement by the presence/absence of lung pleural linings movement by ultrasound | During assessment with point of care ultrasound (10min)
  Ultrasound placed vertically on the anterior chest of a patient will assess for the presence/absence of the horizontal movement of the two lung pleural linings with respiration.
Localization of endotracheal tube placement by the presence/absence of breath sounds detected by Core-Eko augmented stethoscope | During assessment with Core-Eko augmented stethoscope auscultation (5min)
  Presence of breath sounds will be assessed and recorded using Core-Eko augmented stethoscope, in conjunction with the smartphone interface over Bluetooth, by auscultating patient's chest. The technology will display breath sounds as a visual soundwave on the smartphone.
  As a result, this will be used to determine location of endotracheal tube (for example, if breath sounds absent in the left lung, we would infer that the tube is in the right bronchus).

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, MD, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kollef MH, Legare EJ, Damiano M. Endotracheal tube misplacement: incidence, risk factors, and impact of a quality improvement program. South Med J. 1994 Feb;87(2):248-54. doi: 10.1097/00007611-199402000-00020. PMID 8115893
- [Background] Kerrey BT, Rinderknecht AS, Geis GL, Nigrovic LE, Mittiga MR. Rapid sequence intubation for pediatric emergency patients: higher frequency of failed attempts and adverse effects found by video review. Ann Emerg Med. 2012 Sep;60(3):251-9. doi: 10.1016/j.annemergmed.2012.02.013. Epub 2012 Mar 15. PMID 22424653
- [Background] Jemmett ME, Kendal KM, Fourre MW, Burton JH. Unrecognized misplacement of endotracheal tubes in a mixed urban to rural emergency medical services setting. Acad Emerg Med. 2003 Sep;10(9):961-5. doi: 10.1111/j.1553-2712.2003.tb00652.x. PMID 12957980
- [Background] Bissinger U, Lenz G, Kuhn W. Unrecognized endobronchial intubation of emergency patients. Ann Emerg Med. 1989 Aug;18(8):853-5. doi: 10.1016/s0196-0644(89)80211-2. PMID 2757282
- [Background] Geisser W, Maybauer DM, Wolff H, Pfenninger E, Maybauer MO. Radiological validation of tracheal tube insertion depth in out-of-hospital and in-hospital emergency patients. Anaesthesia. 2009 Sep;64(9):973-7. doi: 10.1111/j.1365-2044.2009.06007.x. PMID 19686482
- [Background] Brunel W, Coleman DL, Schwartz DE, Peper E, Cohen NH. Assessment of routine chest roentgenograms and the physical examination to confirm endotracheal tube position. Chest. 1989 Nov;96(5):1043-5. doi: 10.1378/chest.96.5.1043. PMID 2509149
- [Background] Sivit CJ, Taylor GA, Hauser GJ, Pollack MM, Bulas DI, Guion CJ, Fearon T. Efficacy of chest radiography in pediatric intensive care. AJR Am J Roentgenol. 1989 Mar;152(3):575-7. doi: 10.2214/ajr.152.3.575. PMID 2783812
- [Background] Dietrich KA, Strauss RH, Cabalka AK, Zimmerman JJ, Scanlan KA. Use of flexible fiberoptic endoscopy for determination of endotracheal tube position in the pediatric patient. Crit Care Med. 1988 Sep;16(9):884-7. doi: 10.1097/00003246-198809000-00013. PMID 3402233
- [Background] Ramsingh D, Frank E, Haughton R, Schilling J, Gimenez KM, Banh E, Rinehart J, Cannesson M. Auscultation versus Point-of-care Ultrasound to Determine Endotracheal versus Bronchial Intubation: A Diagnostic Accuracy Study. Anesthesiology. 2016 May;124(5):1012-20. doi: 10.1097/ALN.0000000000001073. PMID 26950708
- [Background] Behere S, Baffa JM, Penfil S, Slamon N. Real-World Evaluation of the Eko Electronic Teleauscultation System. Pediatr Cardiol. 2019 Jan;40(1):154-160. doi: 10.1007/s00246-018-1972-y. Epub 2018 Aug 31. PMID 30171267